CLINICAL TRIAL: NCT00001097
Title: Establishment and Maintenance of Long-Term Undetectable Plasma HIV-1 RNA: Correlation With Immunologic Reconstitution and Viral Dynamics
Brief Title: Long-Term Effects of HAART in Youth With Stronger Immune Systems Versus Youth With Weaker Immune Systems
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: ACTG 381; PACTG 381
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to see if children and young adults with better immune systems before starting highly active antiretroviral therapy (HAART) do better than those who have weaker immune systems before starting HAART.

HIV infection weakens the immune system's ability to fight other infections and diseases. HAART is a type of anti-HIV therapy shown to improve the immune system of adults. However, not all patients show the same amount of improvement with HAART. Doctors believe that results may depend on how strong a patient's immune system is before starting HAART. Long-term effects of HAART in children and young adults have not yet been studied.

DETAILED DESCRIPTION:
Recent adult clinical trials involving combination HAART, including a protease inhibitor (PI), have demonstrated improvements in somatic immune system functioning. [AS PER AMENDMENT 2/27/01: More recently, similar success has been demonstrated with a PI-sparing regimen, zidovudine, lamivudine, and efavirenz.] Not all individuals, however, experience the same level of immune reconstitution, and oftentimes any improvement is short-lived. Adolescent patients may have a greater potential for immune restoration because of residual thymic tissue and therefore may experience greater long-term virus-free states as compared to adult patients. This study examines the duration of virologic efficacy HAART has on the adolescent HIV-positive population.

Patients begin study by initiating a HAART regimen of a minimum of 3 drugs, at least 1 of which must be a PI [AS PER AMENDMENT 2/27/01: or efavirenz (EFV)]. A variety of drug combinations are used; therefore, patients are grouped according to the classes of drugs in their respective regimen (e.g., 2 nucleoside reverse transcriptase inhibitors [NRTIs] plus 1 PI; 2 NRTIs plus 2 PIs; 1 or 2 NRTIs plus 1 PI plus 1 nonnucleoside reverse transcriptase inhibitor [NNRTI] [AS PER AMENDMENT 2/27/01: ; and 2 NRTIs plus EFV]). At the time of HAART initiation, patients undergo immunologic and virologic assessments in order to determine baseline values. Then, to determine the virologic success or failure of HAART, HIV-1 RNA measurements are taken and compared to initial baseline values. Virologic success equals undetectable HIV-1 RNA at Week 12 [AS PER AMENDMENT 2/27/01: and confirmed at Week 16] or a significant (greater than 1 log) decrease in HIV-1 RNA from baseline to Week 12 [AS PER AMENDMENT 2/27/01: and confirmed undetectable HIV-1 RNA before the next scheduled visit (Week 24)]. Patients are followed for a minimum of 3 years of maintained viral suppression or until they have demonstrated virologic failure. From these values, any correlation that may exist between HIV-1 RNA values and HAART can be deduced. Patients with virologic failure on the initial HAART regimen may be allowed to change to a second HAART regimen. [AS PER AMENDMENT 2/27/01: Patients with virologic success on the second HAART regimen are followed for a minimum of 3 years.] Patients with virologic failure on the second HAART regimen or who voluntarily discontinue HAART are followed using an abbreviated schedule for 3 years.

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive.
* Are between 8 and 22 years old (consent of parent or guardian required if under 18).
* Have detectable levels of HIV in the blood within 30 days prior to study entry.
* Expect to be on the study for at least 1 year. (This study has been changed by adding this requirement.)
* Are pregnant and are not taking didanosine/stavudine (ddI/d4T) or EFV as part of their HAART regimen. (This study has been changed so that pregnant patients may be eligible if they are not taking ddI/d4T or EFV.)

Exclusion Criteria

Children will not be eligible for this study if they:

* Are taking HAART or more than 1 anti-HIV drug.
* Were infected with HIV before birth, at the time of delivery, or by a blood transfusion during birth.
* Have taken part in the study before.
* Have not responded well to HAART in the past.
* Have taken drugs to boost the immune system such as HIV vaccines, IVIG, or cytokine therapy.
* Have AIDS-related (opportunistic) infection at the time of screening. (This study has been changed so that patients with an AIDS-related infection are ineligible.)
* Are pregnant and are taking ddI/d4T or EFV as part of their HAART regimen. (This study has been changed so that pregnant patients are ineligible if they are taking ddI/d4T or EFV.)

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Flynn, Study Chair
Locations (46):
- United States (43):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - Phoenix Childrens Hosp, Phoenix, Arizona
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Denver, Denver, Colorado
  - Connecticut Children's Med Ctr, Farmington, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Earl K Long Early Intervention Clinic, New Orleans, Louisiana
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Flynn P, Douglas S, Rudy B, Lathey J, Lindsey J, Wang Y. Establishment and maintenance of long-term undetectable plasma HIV-1 RNA: correlation with immunologic reconstitution and viral dynamics. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 692)
- [Result] Wu H, Lathey J, Ruan P, Douglas SD, Spector SA, Lindsey J, Hughes MD, Rudy BJ, Flynn PM; PACTG 381 Team. Relationship of plasma HIV-1 RNA dynamics to baseline factors and virological responses to highly active antiretroviral therapy in adolescents (aged 12-22 years) infected through high-risk behavior. J Infect Dis. 2004 Feb 15;189(4):593-601. doi: 10.1086/381500. Epub 2004 Jan 29. PMID 14767811
- [Result] Flynn PM, Rudy BJ, Douglas SD, Lathey J, Spector SA, Martinez J, Silio M, Belzer M, Friedman L, D'Angelo L, McNamara J, Hodge J, Hughes MD, Lindsey JC; Pediatric AIDS Clinical Trial Group 381 Study Team. Virologic and immunologic outcomes after 24 weeks in HIV type 1-infected adolescents receiving highly active antiretroviral therapy. J Infect Dis. 2004 Jul 15;190(2):271-9. doi: 10.1086/421521. Epub 2004 Jun 18. PMID 15216461
- [Result] Rudy BJ, Lindsey JC, Flynn PM, Bosch RJ, Wilson CM, Hughes ME, Douglas SD; Pediatric Aids Clinical Trials Group 381 Study Team. Immune reconstitution and predictors of virologic failure in adolescents infected through risk behaviors and initiating HAART: week 60 results from the PACTG 381 cohort. AIDS Res Hum Retroviruses. 2006 Mar;22(3):213-21. doi: 10.1089/aid.2006.22.213. PMID 16545007
- [Result] Flynn PM, Rudy BJ, Lindsey JC, Douglas SD, Lathey J, Spector SA, Martinez J, Silio M, Belzer M, Friedman L, D'Angelo L, Smith E, Hodge J, Hughes MD; PACTG 381 Study Team. Long-term observation of adolescents initiating HAART therapy: three-year follow-up. AIDS Res Hum Retroviruses. 2007 Oct;23(10):1208-14. doi: 10.1089/aid.2006.0290. PMID 17961106